CLINICAL TRIAL: NCT00131404
Title: A 2-Year Study to Assess the Efficacy, Safety, and Tolerability of Taranabant in Obese Patients Followed by a 1-Year Extension
Brief Title: A Two Year Safety and Efficacy Study in Obese Patients (0364-015)(TERMINATED)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The overall profile does not support development for obesity
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0364-015; 2005_031
Record Dates: First submitted 2005-08-16; First posted 2005-08-18 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — N-(3-(4-chlorophenyl)-2-(3-cyanophenyl)-1-methylpropyl)-2-methyl-2-((5-(trifluoromethyl)pyridin-2-yl)oxy)propanamide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Phase A/B: Arm 1 (Placebo Comparator): Phase A: Arm 1: MK0364 Pbo capsule once daily.
  Phase B: Patients who continue into Phase B will remain in the same arm they were assigned to during Phase A and will receive the following: Arm 1: MK0364 Pbo capsule once daily.
  Interventions: Drug: Comparator: Placebo
- Phase A/B: Arm 2 (Experimental): Phase A: Arm 2: MK0364 2 mg capsule once daily.
  Phase B: Patients who continue into Phase B will remain in the same arm they were assigned to during Phase A and will receive the following: Arm 2: MK0364 2 mg capsule once daily.
  Interventions: Drug: taranabant
- Phase A/B: Arm 3 (Experimental): Phase A: Arm 3: MK0364 4 mg capsule once daily.
  Phase B: Patients who continue into Phase B will remain in the same arm they were assigned to during Phase A and will receive the following: Arm 3:
  MK0364 4 mg capsule once daily.
  Interventions: Drug: taranabant
- Phase A/B: Arm 4 (Experimental): Phase A: Arm 4: MK0364 6 mg capsule once daily.
  Phase B: Patients who continue into Phase B will remain in the same arm they were assigned to during Phase A and will receive the following: Arm 4:
  MK0364 6 mg capsule once daily.
  Interventions: Drug: taranabant
- Phase A/B: Arm 5 (Experimental): Phase A: Arm 5: MK0364 6 mg capsule once daily. 52 week treatment period. Phase B: Patients who continue into Phase B will remain in the same arm they were assigned to during Phase A and will receive the following: Arm 5: MK0364 6 mg capsule once daily.
  Interventions: Drug: taranabant

INTERVENTIONS:
Drug: taranabant — taranabant 2 mg capsule, 4 mg capsule, 6 mg capsule once daily. 52 week treatment period.
  Other Names: MK0364
  Arms: Phase A/B: Arm 2; Phase A/B: Arm 3; Phase A/B: Arm 4; Phase A/B: Arm 5
Drug: Comparator: Placebo — Placebo capsule once daily. 52 week treatment period.
  Arms: Phase A/B: Arm 1

SUMMARY:
A study to determine the safety and efficacy of an investigational drug in patients with obesity plus extension.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients with a body mass index between 30 kg/m2 and 43 kg/m2, inclusive (BMI between 27 kg/m2 and 43 kg/m2, inclusive for those with obesity-related comorbidities including hypertension, dyslipidemia, and sleep apnea

Exclusion Criteria:

* Patients with serious or unstable current or past medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Actual)
Dates: Start 2005-09; Primary Completion 2007-02 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Decreases body weight; safety and tolerability | 156 Weeks

SECONDARY OUTCOMES:
Decreases waist circumference, the proportion of patients with metabolic syndrome, triglycerides, non-HDL-C, LDL-C, fasting insulin, FPG; increases HDL-C, insulin sensitivity | 156 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Aronne LJ, Tonstad S, Moreno M, Gantz I, Erondu N, Suryawanshi S, Molony C, Sieberts S, Nayee J, Meehan AG, Shapiro D, Heymsfield SB, Kaufman KD, Amatruda JM. A clinical trial assessing the safety and efficacy of taranabant, a CB1R inverse agonist, in obese and overweight patients: a high-dose study. Int J Obes (Lond). 2010 May;34(5):919-35. doi: 10.1038/ijo.2010.21. Epub 2010 Feb 16. PMID 20157323